CLINICAL TRIAL: NCT02010554
Title: Development of a Talk Therapy Protocol to Help Patients Make Treatment Decisions in MS
Acronym: MIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri, Kansas City (Other)
Responsible Party: Principal Investigator, Jared Bruce, Associate Professor of Psychology, University of Missouri, Kansas City
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HC 0138-02; 0033769 (Other Grant/Funding Number: National MS Society)
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-11

CONDITIONS: Relapsing-remitting Multiple Sclerosis
Keywords: Multiple Sclerosis; Disease modifying medication; Relapsing-Remitting MS; Motivational Interviewing; Telephone Counseling
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Brief Education (Active Comparator): Patients receive a brief educational packet along with treatment as usual
  Interventions: Behavioral: Brief Education
- MI-CBT Treatment (Experimental): Patients receive five 20 minute phone sessions of motivational interviewing/cognitive behavioral therapy weekly along with a brief educational packet.
  Interventions: Behavioral: Brief Education; Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Brief Education — Give patients a pamphlet discussing pros and cons of disease modifying therapies
Behavioral: Motivational Interviewing-Cognitive Behavioral Therapy — A telephone based talk therapy discussing pros and cons of medication use in MS.
  Arms: MI-CBT Treatment

SUMMARY:
Between 15-20% of MS patients decide not to initiate disease modifying therapies after being diagnosed with MS. For this study, we will develop a telephone-based talk therapy intervention and then conduct a randomized controlled trial. Patients will be assigned to either 5 weekly 20 minute telephone sessions of psychotherapy or a brief education control condition. We hypothesize that patients undergoing phone therapy will be more likely to indicate they are interested in initiating disease modifying medications than patients given brief education and treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of relapsing remitting MS based on established guidelines
* Not taking recommended therapy
* Provider recommendation for DMT use
* At least 18 years of age
* Access to a telephone
* English speaking

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-12; Primary Completion 2015-03 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Adherence Treatment Survey | 10 weeks after enrollment
  Whether the patient indicates if he/she decided to re-initiate disease modifying therapies on a "yes"/"no" question.

SECONDARY OUTCOMES:
Adherence Treatment Survey | 10 weeks after enrollment
  Whether the patient reports that he/she plans to discuss disease modifying therapies with a care provider on a "yes"/"no" question.
Adherence Treatment Survey | 5 weeks after enrollment
  Whether the patient reports that he/she plans to discuss disease modifying therapies with a care provider on a "yes"/"no" question.
Adherence Treatment Survey | 5 weeks after enrollment
  Whether the patient indicates if he/she decided to re-initiate disease modifying therapies on a "yes"/"no" question.

OTHER OUTCOMES:
Motivation/Readiness Questionnaire | 10 weeks after enrollment
  Whether there is increased self-reported motivation to take disease modifying therapies on a 1-10 likert-type scale.
Motivation/Readiness Questionnaire | 5 weeks after enrollment
  Whether there is increased self-reported motivation to take disease modifying therapies on a 1-10 likert-type scale.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Missouri-Kansas City, Kansas City, Missouri
  - Kessler Rehabilitation Institute, West Orange, New Jersey